CLINICAL TRIAL: NCT05897203
Title: Safety, Pharmacokinetics, and Preliminary Efficacy of Herbal Products for the Treatment of Acute Respiratory Viral Infections Including Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) in Uganda; Phase 2A Open Label Clinical Trial
Brief Title: Clinical Trial of Natural Therapeutics for COVID-19 and Other Acute Respiratory Viral Infections
Acronym: CONAT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Makerere University Lung Institute (Unknown); MRC/UVRI and LSHTM Uganda Research Unit (Other); Directorate of Government Analytical Laboratories (Unknown); Makerere University College of Veterinary Medicine, Animal Resources and Bio-security (Unknown); Makerere University Biomedical Research Centre (Unknown); Natural Chemotherapeutics Research Institute (Unknown)
Responsible Party: Principal Investigator, Bruce J Kirenga, Prof, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CONAT
Record Dates: First submitted 2023-05-25; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Acute Respiratory Infection

STUDY DESIGN:
Intervention Model Description: A phase 2A open-label randomized controlled clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Investigational Medicinal product A (IMP A) + Standard of Care (SoC) (Active Comparator): Participants in this arm will receive the both the Investigational medicinal product (IMP A) and the standard of care
  Interventions: Drug: TAZCOV
- Investigational Medicinal product B (IMP B) + Standard of Care (SoC) (Active Comparator): Participants in this arm will receive the both the Investigational medicinal product (IMP B) and the standard of care
  Interventions: Drug: Vidicine
- Standard of care (SoC) (Other): Participants in this arm will receive only the standard of care
  Interventions: Drug: TAZCOV; Drug: Vidicine

INTERVENTIONS:
Drug: TAZCOV — Herbal Syrup
  Arms: Investigational Medicinal product A (IMP A) + Standard of Care (SoC); Standard of care (SoC)
Drug: Vidicine — Herbal Syrup
  Arms: Investigational Medicinal product B (IMP B) + Standard of Care (SoC); Standard of care (SoC)

SUMMARY:
The trial "Safety, Pharmacokinetics and Preliminary Efficacy of herbal products for the treatment of acute respiratory viral infections including SARS-CoV2 in Uganda; Phase 2A Open Label Clinical Trial" is currently being implemented under the Clinical Trials of Natural therapeutics Program. The trial sample size is 510, and the participants include adults (18 years or more) who fulfill the case definitions of acute respiratory infections (ARI), test positive for one of the target respiratory viruses, are negative for TB on GeneXpert; non-pregnant/non-breast-feeding females, have no history of hypersensitivity to any of the investigational products, and have given written consent to participate in the trial.

The overall objective of the trial is to assess the safety, pharmacokinetics and preliminary efficacy of TazCoV and Vidicine for the treatment of acute respiratory viral infections including (SARS-CoV2, RSV and Influenza A/B) in Uganda.

Primary objectives include:

1. To determine the safety and pharmacokinetics of TAZCOV and Vidicine herbal products among adult participants patients with acute respiratory infections including those due to laboratory-confirmed SARS-CoV2, RSV and Influenza A/B
2. To determine the extent of SARS-CoV2, RSV, and Influenza A/B viral clearance among adult participants patients with acute viral respiratory infection treated using TAZCOV and Vidicine
3. To establish time-to-remission of symptoms among participants patients with acute respiratory infections including those due to laboratory-confirmed SARS-CoV2, RSV and Influenza treated with TAZCOV or Vidicine
4. To evaluate disease progression among participants patients with acute respiratory infections including those due to laboratory-confirmed SARS-CoV2, RSV and Influenza treated with TAZCOV or Vidicine The end points include: Solicited and unsolicited side effects (mild, moderate, severe, adverse and serious adverse events), days to viral clearance (RT-PCR negativity) for those with a positive viral test at enrolment and time to presenting symptom resolution. The Pharmacokinetic endpoints include: the maximum concentration of IMP in plasma [Cmax], time taken for the IMP plasma concentration to reach maximum levels [Tmax] and time taken for the concentration of the IMP in the plasma or the total amount in the body to be reduced by 50%.

ELIGIBILITY:
Inclusion Criteria: ALl adults who

* fulfill ARI case definition
* have signs and symptoms of ARI
* test positive for one of the target respiratory viruses (SARS-CoV2, RSV, or Influenza A/B)
* do not have symptoms suggestive of Pulmonary TB i.e cough for more than 2 weeks, drenching night sweats, evening fevers and marked weight loss.
* can provide informed consent or have a surrogate or legally appointed representative to give consent

Exclusion Criteria:

* Severe acute respiratory illness (SARI)-defined as An acute respiratory illness with a history of fever or measured fever of ≥ 38 °C and cough and/or throat with onset within the past 10 days, requiring hospitalization or with SPO2≤92%
* History of hypersensitivity to the investigational product or components therein
* Conditions that may be regarded as contraindications to the investigational medicinal product include known allergic reactions and rashes to any herbal medicines and any untoward reactions to any herbal medications such as bleeding, headaches, high blood pressure, heart failure, seizures, agitation, etc.
* Severe organ impairment (liver, kidney, brain, heart)
* Inability to return for post-discharge follow-up
* Females who are pregnant or intend to become pregnant or are breastfeeding during the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Solicited and unsolicited side effects (mild, moderate, severe, adverse and serious adverse events). | 9 months
  The outcome measures are cumulative incidences of solicited and unsolicited side effects (mild, moderate, severe adverse events) in the study arms
Time to presenting symptom resolution | 14 days
  Will be assessed by time trends in clinical remission of signs and symptoms in the trial arms
Days to viral clearance (RT-PCR negativity) for those with a positive viral test at enrolment | 7 days
  Will be assessed through ascertaining the proportion with negative PCR on days 3, 5 and 7
Progression to severe-critical ARI requiring hospitalization, oxygen therapy and/or mortality | 14 days
  To be measured by ascertaining the proportion progressing to severe ARI requiring hospitalization, oxygen therapy and/or mortality
Time taken for TazCoV and Vidicine plasma concentration to reach maximum levels [Tmax] | 14 days
  To be measured by time to maximum concentration of TazCoV and Vidicine plasma [Tmax]

CONTACTS AND LOCATIONS:
Locations (1):
- Mulago National Referral Hospital, Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other researchers upon reasonable request through the sponsor
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years after trial end